CLINICAL TRIAL: NCT07181564
Title: FUNCTIONAL ENDOSCOPIC NASAL AND SINUS SURGERY AND ANESTHESIA: Study of Hemodynamic Parameters During General Anesthesia Compared to the Surgical Field, as Well as Assessment of Cerebral Ischemia Intraoperatively by Measurement of S100B Protein and Specific Neuronal Enolase (NSE).
Brief Title: Anesthesia Techniques, Neuroprotection and Surgical Field in FESS Under Controlled Hypotension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University General Hospital of Patras (Other)
Responsible Party: Principal Investigator, Sotiria Rizopoulou, Chief Resident Anesthesioogy, University General Hospital of Patras
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 155D0BCB1A1EDDBEE681727C3DAA49; 0000014333 (Other: university of patras)
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Magnesium Sulfate; Remifentanil; S 100beta; S100 Beta Protein, Human; Neuron-Specific Enolase; Brain Ischemia; Sevoflurane Anaesthesia; Propofol/Remifentanil; Ketamine
Keywords: "Anesthesia", "Controlled Hypotension", "FESS", "S100B", "Neuron-Specific Enolase"
MeSH Terms: conditions — Brain Ischemia | interventions — Propofol; Remifentanil; Ketamine; Magnesium Sulfate; Drug Combinations; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The surgeon who rates the surgical field and the investigator responsible for data analysis are blinded to group allocation. The anesthesiologist is aware of the intervention for safety and drug-delivery reasons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1: Propofol-Remifentanil (TIVA) (Active Comparator): Maintenance of general anesthesia with propofol and remifentanil; no ketamine or magnesium administered.
  Interventions: Drug: Propofol / Remifentanil
- Arm 2: Propofol-Remifentanil + Ketamine + Magnesium (TIVA+) (Active Comparator): Maintenance with propofol and remifentanil plus adjunct continuous infusions of ketamine and magnesium.
  Interventions: Drug: Propofol / Remifentanil; Drug: Ketamine + Magnesium sulfate (drug combination)
- Arm 3: Sevoflurane-Remifentanil (Inhalational) (Active Comparator): Maintenance of general anesthesia with sevoflurane and remifentanil; no ketamine or magnesium administered.
  Interventions: Drug: Sevoflurane and Remifentanil
- Arm 4: Sevoflurane-Remifentanil + Ketamine + Magnesium (Inhalational+) (Active Comparator): Maintenance with sevoflurane and remifentanil plus adjunct continuous infusions of ketamine and magnesium.
  Interventions: Drug: Ketamine + Magnesium sulfate (drug combination); Drug: Sevoflurane and Remifentanil

INTERVENTIONS:
Drug: Propofol / Remifentanil — Maintenance of general anesthesia with propofol and remifentanil; no ketamine or magnesium administered.
  Arms: Arm 1: Propofol-Remifentanil (TIVA); Arm 2: Propofol-Remifentanil + Ketamine + Magnesium (TIVA+)
Drug: Ketamine + Magnesium sulfate (drug combination) — Continuous intraoperative infusion per protocol.
  Arms: Arm 2: Propofol-Remifentanil + Ketamine + Magnesium (TIVA+); Arm 4: Sevoflurane-Remifentanil + Ketamine + Magnesium (Inhalational+)
Drug: Sevoflurane and Remifentanil — Continuous intraoperative infusion per protocol.
  Arms: Arm 3: Sevoflurane-Remifentanil (Inhalational); Arm 4: Sevoflurane-Remifentanil + Ketamine + Magnesium (Inhalational+)

SUMMARY:
This prospective, randomized controlled trial investigates the effect of four different anesthetic maintenance techniques on surgical field conditions, hemodynamic stability, and neuroprotection during functional endoscopic sinus surgery (FESS) performed under controlled hypotension. Patients are randomly assigned to receive either total intravenous anesthesia with propofol-remifentanil, propofol-remifentanil with adjunct ketamine and magnesium, sevoflurane-remifentanil, or sevoflurane-remifentanil with adjunct ketamine and magnesium. Primary outcomes include serum biomarkers of neuronal injury (S100B and neuron-specific enolase, NSE) measured perioperatively, as well as surgical field visibility and intraoperative bleeding scores. Secondary outcomes include recovery profile and postoperative pain.

DETAILED DESCRIPTION:
Functional endoscopic sinus surgery (FESS) is commonly performed under controlled hypotension in order to minimize intraoperative bleeding and optimize the surgical field. However, controlled hypotension may pose a risk of cerebral hypoperfusion and neuronal injury. This prospective, single-center randomized controlled study aims to compare four anesthetic maintenance regimens: (1) propofol-remifentanil, (2) propofol-remifentanil plus continuous ketamine and magnesium infusion, (3) sevoflurane-remifentanil, and (4) sevoflurane-remifentanil plus continuous ketamine and magnesium infusion.

The primary objectives are to evaluate differences in serum S100B and NSE levels at three perioperative time points (baseline before incision, 20 minutes after initiation of controlled hypotension, and at the end of surgery), as well as surgical field quality (7-point Likert scale) and intraoperative bleeding (0-5 scale) as rated by blinded surgeons. Secondary objectives include assessment of extubation conditions with the Aldrete score and evaluation of postoperative pain using a visual analogue scale (VAS). The findings of this trial may help determine whether adjunct agents with potential neuroprotective properties, such as ketamine and magnesium, provide additional benefit during FESS under controlled hypotension.

ELIGIBILITY:
Inclusion Criteria :

Adult patients (≥18 years old). Scheduled for F.E.S.S (Functional endoscopic sinus surgery ) under general anesthesia.

Able to provide informed consent

Exclusion Criteria:

Emergency surgery. ASA physical status IV-V. Severe hepatic or renal dysfunction. Known allergy or contraindication to study drugs. Pregnant or lactating women. unable to provide informed consent

Patients unwilling or unable to provide consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Measure: Serum S100B concentration | Prior to surgical incision (baseline), 20 minutes after initiation of controlled hypotension, and at the end of functional endoscopic sinus surgery (FESS) under controlled hypotension
  S100B measured in blood samples using institutional clinical laboratory immunoassay methods; values reported in standard laboratory units (e.g., ng/mL).
Measure: Serum neuron-specific enolase (NSE) concentration | Prior to surgical incision (baseline), 20 minutes after initiation of controlled hypotension, and at the end of functional endoscopic sinus surgery (FESS) under controlled hypotension
  NSE measured in blood samples using institutional clinical laboratory immunoassay methods; values reported in standard laboratory units (e.g., ng/mL).
Measure: Surgical field quality score (7-point Likert scale) | At the end of surgery
  The blinded surgeon will rate surgical field conditions (visibility and bleeding) on a standardized 7-point Likert scale (1 = severe bleeding, 7 = optimal conditions).
Measure: Intraoperative bleeding score (0-5 scale) | At the end of surgery
  Bleeding during surgery assessed on a 0-5 scale, where higher scores indicate heavier bleeding.

SECONDARY OUTCOMES:
Measure: Extubation conditions (Aldrete score, SAS score) | Immediately after extubation in the operating room / upon PACU arrival
  Recovery profile assessed with the Aldrete score (0-10), evaluating activity, respiration, circulation, consciousness, and SpO₂.
Postoperative pain (VAS 0-10) | Within the first 24 hours postoperatively
  Pain intensity measured using the visual analogue scale (VAS, 0-10). Administration of pethidine (0.5-1 mg/kg IM or IV) will be recorded if analgesia was required.

CONTACTS AND LOCATIONS:
Locations (1):
- University General Hospital of Patras, Pátrai, Achaia, Greece

IPD SHARING:
Plan to Share IPD: No